CLINICAL TRIAL: NCT04016428
Title: Online Prenatal Trial in Mindfulness Sleep Management
Acronym: OPTIMISM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Ira Kantrowitz-Gordon, Assistant Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00005267; 5P30NR016585-02 (NIH)
Record Dates: First submitted 2019-06-18; First posted 2019-07-11 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Pregnancy Related; Insomnia; Depression
Keywords: sleep; pregnancy; insomnia; depression; mindfulness
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OPTIMISM Intervention (Experimental): Participants will receive online delivery of a mindfulness-based program for improving sleep in pregnancy, along with the usual care they would receive from their provider.
  Interventions: Behavioral: OPTIMISM
- Sleep Education (Active Comparator): Participants will receive online delivery of an education program on sleep in pregnancy, along with the usual care they would receive from their provider.
  Interventions: Behavioral: Sleep Education

INTERVENTIONS:
Behavioral: OPTIMISM — Six-week online program that emphasizes mindfulness and skills for improving sleep during pregnancy.
  Arms: OPTIMISM Intervention
Behavioral: Sleep Education — Six-week online program that provides education on sleep during pregnancy.
  Arms: Sleep Education

SUMMARY:
The aim of this study is to assess an online mindfulness intervention for pregnant women (6 weeks) for the treatment of insomnia and prevention of depression relapse in pregnancy. This mindfulness intervention will also be compared with an online intervention (6 weeks) consisting only of education about insomnia in pregnancy. The principal hypothesis is that the mindfulness intervention will be more effective than the education-only intervention.

DETAILED DESCRIPTION:
The aim of this study is to assess an online mindfulness intervention for pregnant women (6 weeks) for the treatment of insomnia and prevention of depression relapse in pregnancy.

There will be two groups:

1. An online mindfulness intervention for pregnant women (6 weeks) that focuses on behaviors to overcome sleep difficulties in pregnancy.
2. An online control group that will receive information about sleep in pregnancy (6 weeks).

Each group will be composed of 25 participants with a total sample of 50. The principal hypothesis is that the mindfulness intervention will be more effective than sleep education in the improvement of sleep and depression symptoms during pregnancy.

The differences between the intervention and control group will be analyzed. The acceptability and usability of online content will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

1) Viable pregnancy in second trimester (up to 28 weeks gestation); 2) prior diagnosis of depression currently in remission (score < 3 on the Patient Health Questionnaire (PHQ-2) depression screening questionnaire); 3) subjective report of insomnia (score > 7 on the Insomnia Severity Index); 4) age 18 or older; 5) access to an Internet-enabled smartphone, tablet, or computer; and 6) English fluency. Participants will not be excluded from participation if they are currently receiving psychotropic medications or psychotherapy.

Exclusion Criteria:

1) Known severe congenital fetal anomalies, fetal demise, or expected neonatal death; 2) diagnosis of major depressive disorder within past 2 months; 3) other significant psychiatric illness requiring treatment; 4) current hospitalization; 5) prior diagnosis of obstructive sleep apnea or restless leg syndrome; 6) positive self-report screen for restless leg syndrome; 7) regular mindfulness or meditative practice (at least weekly); and 8) regular night-shift work.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | Enrollment to intervention completion (6 weeks)
  Self-rating of overall sleep quality and disturbances using 7 sleep components. Total scores range from 0 to 21, with higher scores indicating worse sleep quality. PSQI global >5 is highly sensitive and specific for distinguishing good and poor sleepers. A lower PSQI score is a better outcome.

SECONDARY OUTCOMES:
Sleep efficiency | Enrollment to intervention completion (6 weeks)
  Sleep efficiency will be calculated from total sleep time divided by time in bed, as measured by 8 days of wrist actigraphy and sleep diaries. Increased sleep efficiency is a better outcome.
Total wake time | Enrollment to intervention completion (6 weeks)
  Total wake time will include all time spent in bed awake, measured in minutes. This will be measured by actigraphy and sleep diaries, and will be calculated as the sum of sleep onset latency (time from getting into bed to falling asleep) and wake after sleep onset (time awake after sleep onset). Decreased total wake time is a better outcome.
Total sleep time | Enrollment to intervention completion (6 weeks)
  Total sleep time is the sum of all time spent asleep, measured in minutes. This will be measured by actigraphy and sleep diaries, and calculated as the difference between time in bed and total wake time. Increased total sleep time is a better outcome.
Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance Short Form | Enrollment to intervention completion (6 weeks)
  A six-item self-report questionnaire that measures perception of the quality of sleep over the past seven days. Total score ranges from 6 to 30, with higher scores indicating more disturbed sleep. Decreased sleep disturbance is a better outcome.
PROMIS Sleep-Related Impairment Short Form | Enrollment to intervention completion (6 weeks)
  An eight-item self-report questionnaire for perceptions of alertness, sleepiness, and tiredness during usual waking hours, and the perceived functional impairments during wakefulness associated with sleep problems or impaired alertness. Total scores range from 8 to 40, with higher scores indicating increased impairment over the past 7 days. Decreased impairment is a better outcome.
PROMIS Fatigue Short Form | Enrollment to intervention completion (6 weeks)
  A six-item self-report questionnaire for reporting subjective feelings of tiredness and the impact on the ability to function normally over the past seven days. Total scores range from 6 to 30, with higher scores indicating increased fatigue. Decreased fatigue is a better outcome.
Edinburgh Postnatal Depression Scale (EPDS) | Enrollment to intervention completion (6 weeks)
  A ten-item self-report questionnaire for depression symptoms in the past week validated for use during pregnancy and postpartum. Total scores range from 0 to 30, with higher scores indicating increased symptoms of depression. Decreased depression is a better outcome.
PROMIS Depression Short Form | Enrollment to intervention completion (6 weeks)
  A six-item self-report questionnaire for depression symptoms in the past week. Total scores range from 6 to 30, with higher scores indicating increased symptoms of depression. Decreased depression is a better outcome.
PROMIS Anxiety Short Form | Enrollment to intervention completion (6 weeks)
  A six-item self-report questionnaire for anxiety symptoms in the past week. Total scores range from 6 to 30, with higher scores indicating increased symptoms of anxiety. Decreased anxiety is a better outcome.
Neuro-QOL Positive Affect and Well-Being Short Form | Enrollment to intervention completion (6 weeks)
  A nine-item self-report questionnaire for recent frequency of positive emotions. Total scores range from 9 to 45, with higher scores indicating increased positive emotions. A higher score is a better outcome.
Short Form (36) Health Survey | Enrollment to intervention completion (6 weeks)
  A 36-item, patient-reported survey of patient health status and quality of life. Total scores range from 0 to 100, with lower scores indicating increased disability. Increased scores are a better outcome.
Intervention adherence | Intervention completion (6 weeks)
  Intervention adherence will be measured as the number of intervention modules completed, with a range of 0 to 6. Increased modules completed indicates greater intervention adherence and is a better outcome.
Meditation adherence | Intervention completion (6 weeks)
  Meditation adherence will be measured by the average number of days per week the participant practiced at least one meditation, with a range of 0 to 7. Increased meditation adherence is a better outcome.
Intervention acceptability | Intervention completion (6 weeks)
  Acceptability will be measured by a self-report 8-item questionnaire on program satisfaction, utility, and ease of use. The range of total scores is 8 to 40, with higher scores indicating increased acceptability. Higher acceptability is a better outcome.

OTHER OUTCOMES:
PROMIS Self-Efficacy for Managing Emotions -- Short Form | Enrollment to intervention completion (6 weeks)
  A four-item self-report questionnaire for measuring confidence in handling emotions. Total scores range from 4 to 20, with higher scores indicated greater ability to handle emotions. Increased confidence is a better outcome.
Index of Self-Regulation (ISR) | Enrollment to intervention completion (6 weeks)
  A nine-item self-report questionnaire designed to measure individuals' level of motivation and self-regulation for health-related behavior change. Total scores range from 6 to 54, with higher scores indicating greater self-regulation. Increased self-regulation is a better outcome.
Sleep Problem Acceptance Questionnaire (SPAQ) | Enrollment to intervention completion (6 weeks)
  An 8-item self-report questionnaire that assesses acceptance of insomnia. Total scores range from 0 to 48, with higher scores indicating a higher level of acceptance. Increased acceptance is a better outcome.
Five Facet Mindfulness Questionnaire Short Form (FFMQ-SF) | Enrollment to intervention completion (6 weeks)
  A 24-item self-report questionnaire that measures the trait-like tendency to be mindful in daily life. It includes five subscales, measuring different aspects of mindfulness. Four of the subscale scores range from 5 to 25; one subscale ("observing") has a range of 4 to 20. Higher scores indicate increased mindfulness, which is a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ira Kantrowitz-Gordon, PhD, CNM, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared via the Common Data Repository for Nursing Science (cdRNS) at the National Institute of Nursing Research.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data will become available 6 months after study start-up and will continue to be available throughout the study.
Access Criteria: Steps to access data are available at https://cdrns.nih.gov/access-data

REFERENCES:
- [Derived] Wi D, Lee RY, Kantrowitz-Gordon I. Efficacy of online mindfulness for the treatment of insomnia in pregnancy: A randomized clinical trial. PLoS One. 2025 May 9;20(5):e0322931. doi: 10.1371/journal.pone.0322931. eCollection 2025. PMID 40343904
- [Derived] Kantrowitz-Gordon I, McCurry SM, Landis CA, Lee R, Wi D. Online prenatal trial in mindfulness sleep management (OPTIMISM): protocol for a pilot randomized controlled trial. Pilot Feasibility Stud. 2020 Sep 14;6:128. doi: 10.1186/s40814-020-00675-1. eCollection 2020. PMID 32944276